CLINICAL TRIAL: NCT01249794
Title: Effectiveness of Continuous Positive Airway Pressure Outside the Intensive Care Unit After Cardiac Surgery
Brief Title: Non Invasive Ventilation After Cardiac Surgery
Acronym: CPAP-CCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO/URC/ER/mm 183/DG
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Respiratory Failure
Keywords: NIV; non invasive ventilation; cardiac surgery; continuous positive airway pressure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

ARMS (2):
- Best available treatment (No Intervention)
- non invasive ventilation (Experimental)
  Interventions: Procedure: non invasive ventilation

INTERVENTIONS:
Procedure: non invasive ventilation — continuous positive airways pressure
  Other Names: NIV; CPAP
  Arms: non invasive ventilation

SUMMARY:
Patients with respiratory failure following cardiac surgery are randomized to receive standard therapy versus non invasive ventilation. The hypothesis is that patients receiving non invasive ventilation will perform better than those who received standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* hypoxia

Exclusion Criteria:

* pneumothorax
* cardiocirculatory instability
* no written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ottavio Alfieri, MD, Principal Investigator — Vita-Salute San Raffaele, Milano, Italia
Locations (1):
- Ospedale San Raffaele di Milano, Italy, Milan, Italy